CLINICAL TRIAL: NCT04293536
Title: Incidence of a Retained Surgical Device in Patients That Underwent Surgery
Brief Title: Incidence of Retained Surgical Devices and Treatment
Status: Completed | Type: Observational
Sponsor: Assuta Medical Center (Other)
Responsible Party: Principal Investigator, Sergio Gabriel Susmallian, Medicine Doctor, Assuta Medical Center
Other Study IDs: AMC 1-2020
Record Dates: First submitted 2020-02-29; First posted 2020-03-03 (Actual); Last update posted 2020-03-09 (Actual); Status verified 2020-03

CONDITIONS: Postoperative Complications, Surgical Sponges, Surgical Instruments, Retained Surgical Tools
MeSH Terms: conditions — Postoperative Complications; Foreign Bodies

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Cases study — Patients with a retained device or almost
  Other Names: retained devices

SUMMARY:
It has been estimated that in the United States alone 48 million operations are performed annually and most involve the use of multiple surgical items, including needles and other sharp objects, surgical sponges, and surgical instruments1. Textile material and instruments forgotten in a patient undergoing an invasive procedure is a negligence of an entire team responsible for maintaining patient safety. A retained surgical foreign body (RSFB) usually requires at least a second surgery for retrieval of the object, and also carries a risk for major complications including morbidity and death2. Retained foreign bodies are underreported to minimize exposure to possible litigation3. Therefore, the real occurrence of RSFB is underestimated, recently there has reported an incidence of 0.356 / 1,000 patients whereas others reported a rate of 1/5000 with an associated mortality ranging from 11 to 35% 4-5.

Therefore, there is a need for improved systems and methods for identifying and tracking surgical items, including needles and other sharp objects, surgical sponges, and surgical instruments during a surgical procedure.

DETAILED DESCRIPTION:
All cases investigated due to retained material during hospital surgical treatment will be included. Incidence, type of procedure performed, the prevalence and guilty of the personal actuating will be considered.

ELIGIBILITY:
Inclusion Criteria:

* Any patient who during internment for surgery had an accident of forgetfulness in the material used for their treatment.

Exclusion Criteria:

* No exclusion criteria

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who were admitted to carrying out an intervention in which material used for their treatment was forgotten or almost.
Sampling Method: Non-Probability Sample
Enrollment: 148 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Incidence of retained devices | three years
  Cases with retained devices or almost accident will be considered

SECONDARY OUTCOMES:
Type of devices | 3 years
  Sponge , instruments and others devices

CONTACTS AND LOCATIONS:
Overall Officials: Sergio Susmallian, MD, Principal Investigator — Assuta Medical Center
Locations (2):
- Israel (2):
  - ASSUTAMC, Tel Aviv
  - Assuta MC, Tel Aviv

REFERENCES:
- [Background] Lauwers PR, Van Hee RH. Intraperitoneal gossypibomas: the need to count sponges. World J Surg. 2000 May;24(5):521-7. doi: 10.1007/s002689910084. PMID 10787070
- [Result] Hall MJ, Schwartzman A, Zhang J, Liu X. Ambulatory Surgery Data From Hospitals and Ambulatory Surgery Centers: United States, 2010. Natl Health Stat Report. 2017 Feb;(102):1-15. PMID 28256998
- [Result] Hariharan D, Lobo DN. Retained surgical sponges, needles and instruments. Ann R Coll Surg Engl. 2013 Mar;95(2):87-92. doi: 10.1308/003588413X13511609957218. PMID 23484986
- [Result] Berkowitz S, Marshall H, Charles A. Retained intra-abdominal surgical instruments: time to use nascent technology? Am Surg. 2007 Nov;73(11):1083-5. PMID 18092638
- [Result] Cima RR, Kollengode A, Garnatz J, Storsveen A, Weisbrod C, Deschamps C. Incidence and characteristics of potential and actual retained foreign object events in surgical patients. J Am Coll Surg. 2008 Jul;207(1):80-7. doi: 10.1016/j.jamcollsurg.2007.12.047. Epub 2008 May 23. PMID 18589366
- [Result] Recommended practices for sponge, sharp, and instrument counts. AORN Recommended Practices Committee. Association of periOperative Registered Nurses. AORN J. 1999 Dec;70(6):1083-9. doi: 10.1016/s0001-2092(06)62224-2. No abstract available. PMID 10635432
- [Result] Steelman VM, Shaw C, Shine L, Hardy-Fairbanks AJ. Retained surgical sponges: a descriptive study of 319 occurrences and contributing factors from 2012 to 2017. Patient Saf Surg. 2018 Jun 29;12:20. doi: 10.1186/s13037-018-0166-0. eCollection 2018. PMID 29988638
- [Result] Brooks J. US Medicare will stop paying for preventable errors. CMAJ. 2007 Oct 9;177(8):841-2. doi: 10.1503/cmaj.071347. No abstract available. PMID 17923647
- [Result] Wan W, Le T, Riskin L, Macario A. Improving safety in the operating room: a systematic literature review of retained surgical sponges. Curr Opin Anaesthesiol. 2009 Apr;22(2):207-14. doi: 10.1097/ACO.0b013e328324f82d. PMID 19390247
- [Derived] Susmallian S, Folv E, Szyper-Kravitz M. Assessing the diagnostic value of radiographs for retained surgical items: a cautionary analysis. Br J Radiol. 2026 Jan 1;99(1177):150-156. doi: 10.1093/bjr/tqaf241. PMID 41143897
- [Derived] Susmallian S, Barnea R, Azaria B, Szyper-Kravitz M. Addressing the important error of missing surgical items in an operated patient. Isr J Health Policy Res. 2022 Apr 5;11(1):19. doi: 10.1186/s13584-022-00530-z. PMID 35382877